CLINICAL TRIAL: NCT02111603
Title: Ability of Mayo Clinic HPLC Method to Measure Fecal Bile Acids to Demonstrate Response to Colesevelam in Patients With Diarrhea Predominant Irritable Bowel Syndrome
Brief Title: Ability of Mayo Clinic High-performance Liquid Chromatography (HPLC) Method to Measure Fecal Bile Acids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-000384; R01DK092179 (NIH); UL1TR000135 (NIH)
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Diarrhea Predominant Irritable Bowel Syndrome
MeSH Terms: interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Colesevelam (Other): 1875 mg of Colesevelam orally twice daily for 10 days
  Interventions: Drug: Colesevelam

INTERVENTIONS:
Drug: Colesevelam — Subjects will receive 1875 mg of Colesevelam orally twice daily for 10 days
  Other Names: Welchol

SUMMARY:
The investigators' hypothesis is that therapy with Colesevelam, reduces fecal bile acid excretion in patients with Irritable Bowel Syndrome (IBS)-diarrhea with prior evidence of increased fecal 48 hour total bile acid excretion. The investigators aim to study the ability of the HPLC assay for fecal bile acids to demonstrate responsiveness after treatment with Colesevelam.

DETAILED DESCRIPTION:
This study will evaluate whether Colesevelam, a bile acid sequestrant, is able to reduce fecal bile acids and improve bowel function in patients with IBS-diarrhea and Mayo's HPLC method can demonstrate a response to the Colesevelam.

The study design will be a single center, unblinded, single dose trial to study the ability to identify the effect of taking 1875 mg (3 tablets [625 mg/tablet]) of Colesevelam orally twice daily for ten days on fasting serum 7alphaC4 and total 48 hour fecal bile acid excretion. Stool and fasting serum samples will be collected predose and during final 48 hours' dosing for assessment. Participants will also fill out an 8-day stool diary assessing frequency, consistency, ease of passage of bowel movements before and during treatment with Colesevelam.

ELIGIBILITY:
Patients with IBS-diarrhea with prior evidence of increased fecal 48 hour total bile acid and increased fasting serum 7alphaC4 who meet the following:

INCLUSION CRITERIA

* Bowel disease questionnaire (BDQ) - IBS symptoms: Positive by Rome lll criteria
* No restrictions on Hospital Anxiety/Depression Score (HADS).
* Gender: Men or women. Women of childbearing potential will have a negative pregnancy test before initiation of medication.

EXCLUSION CRITERIA

* Use of drugs or agents within the past 1 week or planned use in the subsequent 2 weeks during the study period (Birth control pill, estrogen replacement therapy, and thyroxine replacement are permissible exceptions):

  * Agents that alter GI transit including opioids, narcotics, anticholinergics, tricyclic antidepressants, serotonin-norepinephrine reuptake inhibitors (SNRI) antidepressants.
  * Analgesic drugs including opiates, nonsteroidal anti-inflammatory drugs (NSAID), cyclooxygenase-2 (COX 2) inhibitors
  * Intake of medication that could interfere with the interpretation of the study.
* Female subjects who are pregnant or breast-feeding. Females must be either surgically sterilized, postmenopausal (>12 months since last menses), or, if of childbearing potential, using reliable methods of contraception as determined by the physician.
* Abdominal surgery (except Appendectomy)
* Patients with known chronic liver disease or history of elevated aspartate aminotransferase (AST)/ alanine transaminase (ALT) 2.0 X upper limit of normal.

  * Bile acid (BA) synthesis and possible false positive or negative fecal bile acid or serum 7alpha-hydroxy-4-cholesten-3-one (7alphaC4) result. If there is no AST or ALT values in the medical record, the study physicians will determine if the tests need to be run.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data already published in PMID: 25594801

REFERENCES:
- [Result] Camilleri M, Acosta A, Busciglio I, Boldingh A, Dyer RB, Zinsmeister AR, Lueke A, Gray A, Donato LJ. Effect of colesevelam on faecal bile acids and bowel functions in diarrhoea-predominant irritable bowel syndrome. Aliment Pharmacol Ther. 2015 Mar;41(5):438-48. doi: 10.1111/apt.13065. Epub 2015 Jan 16. PMID 25594801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: 13 subjects were accrued. One subject withdrew from the study after the pre-drug activities, but before the treatment activities.
Period: Overall Study
Arm/Group | Colesevelam
Started | 13
Completed | 12
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 13 subjects were accrued. One subject withdrew from the study after the pre-drug activities, but before the treatment activities.
Arm/Group | Colesevelam
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 12
Mean Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.1 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total 48 Hour Fecal Bile Acids (BA) From Baseline in Response to Treatment With Colesevelam
Description: Stool 48 hour collections (for BAs) were collected during baseline before treatment, and then during days 9-10 of the 10 days of colesevelam dosing for fecal BAs. Total fecal BA were measured using HPLC/tandem mass spectrometry.
Time Frame: baseline, 10 days
Population: 13 subjects were accrued. One subject withdrew from the study after the pre-drug activities, but before the treatment activities. Only the 12 participants with complete data at both baseline and after 10 days of treatment are included in the Outcome Measure.
Measure: Mean (Standard Error); unit: uM
Arm/Group | Colesevelam
Number analyzed (Participants) | 12
uM
  Baseline | 1662 (234.7)
  After 10 days treatment with colesevelam | 3496 (709.2)
Statistical Analysis 1: Comparison: Colesevelam; Comparison of on-treatment total fecal bile acid excretion with baseline total fecal bile acid excretion; Test type: Superiority or Other; p = 0.012, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Fasting Serum C4
Description: Change in fasting serum C4 from baseline in response to treatment with colesevelam.
Time Frame: baseline, 10 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Colesevelam
Number analyzed (Participants) | 12
ng/mL
  Baseline | 24.7 (4.2)
  After 10 days treatment with colesevelam | 72.3 (12.2)

3. Secondary Outcome: Change in Fecal Fat Excretion
Description: Change in fecal fat excretion from baseline in response to treatment with colesevelam
Time Frame: baseline, 10 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/day
Arm/Group | Colesevelam
Number analyzed (Participants) | 12
g/day
  Baseline | 6.4 (1.2)
  After 10 days treatment with colesevelam | 6.8 (0.9)

4. Secondary Outcome: Change in Stool Consistency
Description: The subjects rated their stool consistency using the Bristol Stool Form Scale. The Bristol Stool Form Scale is a medical aid designed to classify the form of human feces into seven categories or types. Types 1 and 2 indicate constipation with 3 and 4 being the "ideal stools" especially the latter, as they are the easiest to defecate, and 5-7 tending towards diarrhea.
Time Frame: baseline, 10 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Colesevelam
Number analyzed (Participants) | 12
units on a scale
  Baseline | 4.8 (0.3)
  After 10 days treatment with colesevelam | 4.4 (0.3)

5. Secondary Outcome: Change in Stool Frequency (Number of Stools Per Week)
Description: Change in stool frequency from baseline in response to treatment with colesevelam.
Time Frame: baseline, 10 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Number of stools per week
Arm/Group | Colesevelam
Number analyzed (Participants) | 12
Number of stools per week
  Baseline | 17.6 (0.4)
  After 10 days treatment with colesevelam | 15.1 (1.9)

6. Secondary Outcome: Concordance Correlation Coefficients of the Relative Composition of Stool Total and the Main Individual Bile Acids (BA)
Description: Stool 48 hour collections (for BAs) were collected during baseline before treatment, and then during days 9-10 of the 10 days of colesevelam dosing for fecal BAs. Relative composition of the main individual bile acids (cholic acid (CA), chenodeoxycholic acid (CDCA), deoxycholic acid (DCA), lithocholic acid (LCA) and ursodeoxycholic acid (UDCA)) in 48 hour stool collection after colesevelam treatment were compared to baseline values.
  The concordance correlation coefficient (rc) measures agreement between two variables. The concordance correlation satisfies -1 ≤ rc ≤ +1. A value of rc = +1 corresponds to perfect agreement. A value of rc = -1 corresponds to perfect negative agreement, and a value of rc = 0 corresponds to no agreement.
Time Frame: baseline, 10 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: concordance correlation coefficient
Arm/Group | Colesevelam
Number analyzed (Participants) | 12
concordance correlation coefficient
  Total BAs at Baseline | 0.53 (0.13)
  Total BAs 48 hour collection after colesevelam | 0.54 (0.15)
  CA at Baseline | 0.84 (0.08)
  CA 48 hour collection after colesevelam | 0.83 (0.06)
  DCA at Baseline | 0.68 (0.14)
  DCA 48 hour collection after colesevelam | 0.85 (0.07)
  UDCA at Baseline | 0.96 (0.20)
  UDCA 48 hour collection after colesevelam | 0.54 (0.20)
  CDCA at Baseline | 0.88 (0.05)
  CDCA 48 hour collection after colesevelam | 0.90 (0.06)
  LCA at Baseline | 0.44 (0.21)
  LCA 48 hour collection after colesevelam | 0.88 (0.07)

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events for the 10 days they were on study.
Arm/Group | Colesevelam
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colesevelam (N=12)
Constipation (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes